CLINICAL TRIAL: NCT06563141
Title: A Suggested Rehabilitation Protocol for the Treatment of C-shape Scoliosis: a Randomized Control Trial
Brief Title: A Suggested Rehabilitation Protocol for the Treatment of C-shape Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khalid safwat elsayed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: khalid-005244
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Scoliosis; Scoliosis Idiopathic; Rehabilitation; C-shape
MeSH Terms: interventions — Traction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traction with mobilization (Experimental): it consists of 35 patients and patients will receive traction with mobilization 3 sessions per week for 3 months with a total of 36 sessions. there will be a follow-up for 2 months with home program exercises and postural instructions only followed by the same pre and post-treatment assessment measures
  Interventions: Other: traction and mobilization
- active exercise therapy) (Active Comparator): it consists of 35 patients and patients will active exercises 3 sessions per week for 3 months with a total of 36 sessions. there will be a follow-up for 2 months with home program exercises and postural instructions only followed by the same pre and post-treatment assessment measures
  Interventions: Other: active exercise therapy

INTERVENTIONS:
Other: traction and mobilization — The patient undergoes a 15-minute infrared therapy session, followed by flexibility and stretching exercises targeting the trunk and four extremities muscles. Land manipulation techniques are used for cervical, dorsal, and lumbar spine to assess and treat spinal dysfunctions. Deep breathing exercises with rib mobilization are also performed to promote respiratory function and thoracic flexibility. The session aims to improve overall health.
  Arms: traction with mobilization
Other: active exercise therapy — Patients with adolescent idiopathic scoliosis will receive exercise programs from seven major schools under SOSORT, focusing on realigning the spine, rib cage, shoulders, and pelvis to normal anatomical postures.
  Arms: active exercise therapy)

SUMMARY:
This study aims to compare the effectiveness of mechanical traction and 3D apical vertebral mobilization and active exercises on Cobb's angle, spinal ROM, and function in patients with C-shaped scoliosis.

DETAILED DESCRIPTION:
Scoliosis is a skeletal issue causing asymmetries, leading to functional disruptions. Common symptoms include uneven eye tilt, drop asloped shoulder, and muscle imbalances. These changes can affect the patient's physical appearance and psychological state. Current treatments have shown suboptimal results due to the lack of accepted scientific theories for idiopathic scoliosis. Therefore, a new therapeutic approach is needed to provide novel insights and improve treatment outcomes. This underscores the need for a more comprehensive approach to scoliosis treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult individuals aged 18 to 30 years (after complete ossification and before the start of the ageing process and joint changes) as mentioned in studies.
2. Thoracolumbar scoliosis with Cobb angle between 10 to 30 degrees because a curve below 10 degrees has no effect and above 30 is indicated for surgery.

Exclusion Criteria:

1. History of orthopaedic surgeries.
2. History of road traffic accidents (RTA).
3. Myopathy.
4. True leg length discrepancy.
5. Neuropathy.
6. Mental disorders.
7. Bone tumor.
8. Heart disease or circulatory problems.
9. Early osteoporosis.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
assessment of degree of spinal curvature | at baseline and after 3 months
  it will be assessed using the scoliometer which is typically consists of a level or inclinometer attached to a base. The scoliometer is placed along the spine, and the angle of deviation from the vertical is measured to assess the severity of the curvature

SECONDARY OUTCOMES:
assessment of the change of the weight, height and body mass index | at baseline and after 3 months
  This scale (DT-150, Shanghai, China) Figure (3) will be used for the measurement of height and weight for each participant and the results will be used for the calculation of the Body Mass Index
assessment of the change of the trunk flexion and extension ROM | at baseline and after 3 months
  To measure flexion, the patient should bend forward at the waist comfortably without knees, and the examiner should stabilize the goniometer's stationary arm on the midline of the spine.
assessment of the change of the trunk lateral flexion ROM | at baseline and after 3 months
  To measure lateral flexion, the patient should lean comfortably sideways without bending forward or rotating the trunk, while the goniometer's stationary arm should be stabilized at the appropriate level.
assessment of the change of the trunk rotation ROM | at baseline and after 3 months
  To measure rotation, the patient rotates their trunk comfortably without moving their hips or feet. The goniometer is placed parallel to the ground, using the scapula's spine as a reference point. The stationary arm remains parallel to the starting position.
assessment of the change of the cervical flexion and extension ROM | at baseline and after 3 months
  To measure flexion, the patient should comfortably lower their chin towards their chest without bending their upper back or shoulders, maintaining straight-forward eyes.
assessment of the change of the cervical lateral flexion ROM | at baseline and after 3 months
  To measure lateral flexion, the patient should tilt their head sideways comfortably without rotating their head or shoulders, keeping their chin level during the movement.
assessment of the change of the cervical rotation ROM | at baseline and after 3 months
  To measure rotation, the patient should comfortably turn their head left or right without tilting their head or shoulders, maintaining straight eyes during the movement.
assessment of the change of fingertips to floor distance | at baseline and after 3 months
  The finger-to-floor distance test is a quick and convenient method to assess hamstring and lower back flexibility. It involves standing up straight, bending forward, lowering hands, reaching the endpoint, and measuring the distance between fingers and the floor.
assessment of the change of the degree of spinal curvature | at baseline and after 3 months
  To measure the Cobb angle on an X-ray, identify the vertebrae with the most tilted endplates, draw lines along the spine's curvature, draw perpendicular lines intersecting at a right angle, and measure the Cobb angle, which represents the degree of spinal curvature.

CONTACTS AND LOCATIONS:
Locations (1):
- May University in Cairo (MUC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No